CLINICAL TRIAL: NCT06497634
Title: Effect of Needle Types and Diameters Using in Spinal Anesthesia on Optic Nerve Sheath Diameter; Prospective Randomized Study
Brief Title: Effect of Spinal Needle Type on Optic Nerve Sheath Diameter
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Sezen Kumaş Solak, Principle Investigator, Bagcilar Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Bagcilar1
Record Dates: First submitted 2024-03-24; First posted 2024-07-12 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Spinal Anesthesia; Intracranial Pressure Change; Optic Nerve Sheath Diameter; Orthopedic Surgery; Cerebrospinal Fluid Leak
MeSH Terms: conditions — Cerebrospinal Fluid Leak

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 25w (25 gauge Whitacre needle) (Active Comparator): Spinal anesthesia will be performed with 25 G pencil point needle (Whitacre)
  Interventions: Procedure: 25 PP; Other: Optic Nerve Sheath Measurement
- Group 25q (25 gauge Quincke needle) (Active Comparator): Spinal anesthesia will be performed with 25 G sharp edge needle (Quincke)
  Interventions: Procedure: 25 Q; Other: Optic Nerve Sheath Measurement
- Group 27q (27 gauge Quincke needle) (Active Comparator): Spinal anesthesia will be performed with 27 G sharp edge needle (Quincke)
  Interventions: Procedure: 27 Q; Other: Optic Nerve Sheath Measurement

INTERVENTIONS:
Procedure: 25 PP — Spinal anesthesia will be performed in sitting position, with 25 G pencil point needle (Whitacre -Egemen®) midline through the L4-5 or L5-S1 interspace, parallel to the dural fibers. Upon clear cerebrospinal fluid (CSF) detection, the needle apertures will be turned towards the cephalad direction, and 3 ml (15 mg) of 0.5% hyperbaric bupivacaine (Marcaine Heavy ®) will be injected into the intrathecal space.
  Arms: Group 25w (25 gauge Whitacre needle)
Procedure: 25 Q — Spinal anesthesia will be performed in sitting position, with 25 G sharp edge needle (Quincke -Egemen®) midline through the L4-5 or L5-S1 interspace, parallel to the dural fibers. Upon clear cerebrospinal fluid (CSF) detection, the needle apertures will be turned towards the cephalad direction, and 3 ml (15 mg) of 0.5% hyperbaric bupivacaine (Marcaine Heavy ®) will be injected into the intrathecal space.
  Arms: Group 25q (25 gauge Quincke needle)
Procedure: 27 Q — Spinal anesthesia will be performed in sitting position, with 27 G sharp edge needle (Quincke -Egemen®) midline through the L4-5 or L5-S1 interspace, parallel to the dural fibers. Upon clear cerebrospinal fluid (CSF) detection, the needle apertures will be turned towards the cephalad direction, and 3 ml (15 mg) of 0.5% hyperbaric bupivacaine (Marcaine Heavy ®) will be injected into the intrathecal space.
  Arms: Group 27q (27 gauge Quincke needle)
Other: Optic Nerve Sheath Measurement — Sonographic measurement of ONSD (EsaoteMyLabFive, Cenova, Italy) for all patients will be performed by a single experienced anesthesiologist. After a thin gel layer apply to the upper eyelid, the patient in the supine position and with the eyes closed, using a 6-13 MHz linear probe, optic sheath nerve measurement will be done 3 mm behind the optic globe, with a total of three measurements of which the final value will be recorded.The measurement will be repeated five times using US guidance at the following time points: T0 (pre-anesthesia), T1 (5 minutes after spinal block), T2 (15 minutes after spinal block, T3 (tourniquet opening), and T4 (24 hours after spinal block ) respectively.

SUMMARY:
The optic nerve sheath is a continuation of the dura mater, extending along the subarachnoid space surrounding the optic nerve. Consequently, changes in intracranial pressure cause an augmentation or contraction in the diameter of the optic nerve sheath, which is coreleted with intracranial pressure. Participants undergoing lower extremity operations (ankle, distal tibia and fibula surgeries) using a tourniquet under spinal anesthesia will be investigated. Spinal anesthesia will be performed with a 25 G Whitacre, 25 G Quincke, or 27 G Quincke needle, depending on the study group. Optic nerve sheath diameter (ONSD) measurements will be performed before spinal anesthesia; and 5 minutes, 15 minutes,,24 hours after spinal block, respectively.The 4th measurement will be performed after tourniquet is opened. Measurements will be done with 15 MHz linear ultrasound (US) probe in B mode, 3 mm behind the posterior globe in the transverse plane from both eyes, on upper eyelid. Values will be recorded numerically. The impact of spinal anesthesia administered using various needle designs (Quincke and Whitacre) and sizes (25G-27G) on intracranial pressure will be investigated.

DETAILED DESCRIPTION:
Optic nerve sheath diameter (ONSD) measured with US emerges as a standout intracranial pressure reflector among non-invasive modalities as a bed side assessment. Different types of needles used in spinal anesthesia cause different lesions in the dura. Lesions created by Quincke needles are small and clean-cut opening in the dural membrane, while those from Whitacre needles result in a more traumatic opening. Also it is known that CSF leakage increase when larger needles are used. As one of postspinal headache mechanism is decrease in the intracranial pressure, the investigators aim to investigate the ONSD changes reflecting intracranial pressure changes.

Participants undergoing lower extremity operations (ankle, distal tibia and fibula surgeries) using a tourniquet under spinal anesthesia will be investigated. Spinal anesthesia will be performed with a 25 G Whitacre, 25 G Quincke, or 27 G Quincke needle, depending on the study group. ONSD measurements will be performed before spinal anesthesia as baseline; and 5 minutes, 15 minutes, 24 hours after spinal block, respectively. Also a measurement will be performed after opening of the surgical tourniquet. Measurements will be done with 15 MHz linear ultrasound (US) probe in B mode, 3 mm behind the posterior globe in the transverse plane from both eyes. Values will be recorded numerically. The impact of spinal anesthesia administered using various needle designs (Quincke and Whitacre) and sizes (25G-27G) on intracranial pressure will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I-II Risk Classification
* Elective orthopedic lower extremity surgery
* Using a tourniquet
* Spinal anesthesia

Exclusion Criteria:

* Bilateral tourniquet usage
* History of orbital trauma
* Optic nerve pathology
* Glaucoma
* Asthma
* Coronary obstructive or pulmonary disease
* Previous corneal or intraocular surgery
* Increased intracranial pressure
* Coagulopathy
* Local site infection
* Refusing to participate in the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 165 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2024-12-25 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Optic nerve sheath diameter | ONSD changes from baseline, at 5 minutes, 15 minutes, 24 hours after spinal anesthesia and opening the tourniquet
  The primary aim is to compare optic nerve sheath diameter (ONSD) according to the spinal needle type and size

SECONDARY OUTCOMES:
Blood pressure | Changes from baseline, at 5 minutes, 15 minutes, 24 hours after spinal anesthesia and opening the tourniquet
  The effect of needle type and size on blood pressure
Hearth rate | Changes from baseline, at 5 minutes, 15 minutes, 24 hours after spinal anesthesia and opening the tourniquet
  The effect of needle type and size on hearth rate
Oxygen saturation | Changes from baseline, at 5 minutes, 15 minutes, 24 hours after spinal anesthesia and opening the tourniquet
  The effect of needle type and size on oxygen saturation

OTHER OUTCOMES:
Nause and vomiting | First 24 hours
  Number of participants with nause and vomiting in first 24 hours
Double vision | First 24 hours
  Number of participants with double vision in first 24 hours
Headache | First 24 hours
  Number of participants with headache in first 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: sezen kumas solak, MD, Principal Investigator — Bagcılar Training Research Hospital
Locations (1):
- Bagcılar Training Research Hospital, Istanbul, Bagci̇lar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The investigators will not share individual patient data

REFERENCES:
- [Background] Reina MA, de Leon-Casasola OA, Lopez A, De Andres J, Martin S, Mora M. An in vitro study of dural lesions produced by 25-gauge Quincke and Whitacre needles evaluated by scanning electron microscopy. Reg Anesth Pain Med. 2000 Jul-Aug;25(4):393-402. doi: 10.1053/rapm.2000.7622. PMID 10925937
- [Background] Killer HE, Laeng HR, Flammer J, Groscurth P. Architecture of arachnoid trabeculae, pillars, and septa in the subarachnoid space of the human optic nerve: anatomy and clinical considerations. Br J Ophthalmol. 2003 Jun;87(6):777-81. doi: 10.1136/bjo.87.6.777. PMID 12770980
- [Background] Tarkkila PJ, Heine H, Tervo RR. Comparison of Sprotte and Quincke needles with respect to post dural puncture headache and backache. Reg Anesth. 1992 Sep-Oct;17(5):283-7. PMID 1419942
- [Derived] Kumas Solak S, Demirgan S, Karali E, Selcan A. Effect of needle types and diameters using in spinal anesthesia on optic nerve sheath diameter: Prospective randomized study. Medicine (Baltimore). 2024 Oct 11;103(41):e40003. doi: 10.1097/MD.0000000000040003. PMID 39465875